CLINICAL TRIAL: NCT04915924
Title: Post Market Surveillance of the HeartMate 3 Left Ventricular Assist System in Korea (Korea HM3 PMS)
Brief Title: Post Market Surveillance of the HeartMate 3 Left Ventricular Assist System in Korea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10344
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Advanced Heart Failure
Keywords: HeartMate 3; ABT-CIP-10344; Left ventricular assist device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HeartMate 3™ left ventricular assist system (HM3 LVAS) (Experimental): Patients will be implanted with the HM3 LVAS
  Interventions: Device: HeartMate 3™ left ventricular assist system (HM3 LVAS)

INTERVENTIONS:
Device: HeartMate 3™ left ventricular assist system (HM3 LVAS) — Advanced heart failure patients will be implanted with the HM3 LVAS

SUMMARY:
The Korea HM3 PMS is a prospective, single arm, open-label, multi-center, post market surveillance is designed to evaluate clinical and functional outcomes with the HM3 LVAS as a treatment for advanced heart failure. The PMS will enroll up to 300 patients, that meet the Health Insurance Review and Assessment (HIRA) guidelines for LVAD implantation, from up to 25 sites in South Korea. Subjects who will be implanted but not included in the PMS can be enrolled retrospectively after obtaining their informed consent. The surveillance period for this PMS is expected to be 4 years from the time of HM3 approval in Korea, concluding on June 2, 2024.

ELIGIBILITY:
Inclusion Criteria

General Inclusion Criteria: All patients approved for HM3 implantation in Korea as per HIRA guidelines will be eligible to be enrolled in the PMS. Only the patients who provide written informed consent will be included in the study. If a subject has had an outcome after the HM3 implantation but prior to providing informed consent, no consent will be obtained, and a limited anonymized data will be collected.

Exclusion Criteria

General Exclusion Criteria: This post market surveillance does not have specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Number of participants with overall survival to transplant, myocardial recovery or on device support free of debilitating stroke (60 days post-stroke Modified Rankin Score >3) or reoperation for pump replacement | Throughout the study (approximately 4 years)
  Overall survival to transplant, myocardial recovery or on device support free of debilitating stroke (60 days post-stroke Modified Rankin Score >3) or reoperation for pump replacement will be assessed using the Kaplan-Meier product-limit method along with a competing outcomes graph. Subjects who are urgently transplanted due to a HeartMate 3 malfunction will be considered to have experienced a primary endpoint event, as will subjects who expire, suffer a debilitating stroke or have their HeartMate 3 exchanged due to a device failure. Subjects who are transplanted (except as described above), explanted for recovery, withdraw from the trial or are lost to follow-up will be censored at that time in the analysis.
Primary Safety Endpoint: Number of cumulative occurrence of adverse events | Throughout the study (approximately 4 years)
  Cumulative occurrence of adverse events will be presented as percent of patients with adverse events and events per patient year of support.

SECONDARY OUTCOMES:
Mean change in Six-minute Walk Test from baseline | Through study completion, an average of 4 years
  The 6-minute Walk test will be conducted at all follow-up visits until the end of the surveillance period. Distance walked at each visit will be compared to baseline using Wilcoxon signed-rank test. To assess the overall changes, repeated measure analysis will be performed using all data collected from baseline to the end of the surveillance period. The overall mean, median, standard deviation, minimum, and maximum will be presented for all follow-up visits. Differences in walking distance between each visit and baseline will be calculated and assessed for improvements using paired, nonparametric Wilcoxon signed-rank test. In addition, box plots will be used to show changes in walking distance over time.
Change in proportion of New York Heart Association (NYHA) Functional Status from baseline | Through study completion, an average of 4 years
  Percent of subjects in each NYHA class will be presented for all follow-up visits. For comparison, patients will be grouped into NYHA Class I/II (No limitation and Slight limitation of physical activity) vs. NYHA Class III/IV (Marked limitation and Inability to carry out physical activities). McNemar's test will be used to assess if there is an increase in proportion of Class I and II subjects at each visit comparing to the baseline.
Mean change in EQ-5D-5L quality of life (QoL) from baseline | Through study completion, an average of 4 years
  Subject's quality of life will be measured by the EQ-5D-5L QoL questionnaire at baseline and all visits after HM3 implant until the end of surveillance period. The overall mean, median, standard deviation, minimum and maximum will be presented for all follow-up visits. Differences in QoL Score between each visit and baseline will be calculated and assessed for improvements using paired, nonparametric Wilcoxon signed-rank test. In addition, box plots will be used to show changes in QoL over time.
Frequency of Rehospitalization and Reoperation | Throughout the study (approximately 4 years)
  Frequency and reason will be reported for rehospitalization and reoperation. Freedom from rehospitalization and reoperation will be assessed using the Kaplan-Meier product-limit method.
Number of participants with Device Malfunctions | Throughout the study (approximately 4 years)
  All suspected HM3 device malfunctions will be reported. Device malfunctions will be collected under the general category of Device Deficiencies. Device deficiency is defined as an inadequacy of a medical device related to its identity, quality, durability, reliability, safety or performance, such as malfunction, misuse or use error and inadequate labeling. This includes the failure of the device to meet its performance specifications or otherwise perform as intended. Data on device malfunctions will be analyzed for the following:
  * The component of the device involved
  * Days to the malfunction
  * Action taken in response to the malfunction
  * Reoperations due to malfunction
  * Death due to malfunction
Incidence of adverse events including, but not limited to, neurological dysfunction, bleeding, infections and device thrombosis. | Throughout the study (approximately 4 years)
  Incidence of adverse events will be assessed including, but not limited to, neurological dysfunction, bleeding, infections and device thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gazzola, Principal Investigator — Abbott
Locations (22):
- South Korea (22):
  - Incheon Sejong Hospital, Incheon, Nam-gu
  - Korea University Ansan Hospital, Ansan
  - Sejong Hospital, Bucheon-si
  - Pusan National University Hospital, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital (CNUH), Gwangju
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong
  - Hallym University Sacred Heart Hospital, Hwaseong
  - Seoul National University Hospital, Ihwa-dong
  - Gachon University Gil Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - St. Mary's Hospital, The Catholic University of Eunpyeong, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No